CLINICAL TRIAL: NCT06344351
Title: A Phase I Study to Evaluate the Safety, Tolerance and Pharmacokinetics of TQB3006 Tablets in Patients With Advanced Malignant Cancer
Brief Title: A Clinical Trial of TQB3006 Tablets in Patients With Advanced Malignant Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3006-I-01
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Advanced Malignant Neoplasm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3006 tablets (Experimental): TQB3006 tables is administered as a single dose or multiple dose .Take200-1200 mg per day; Take TQB3006 orally on an empty stomach once or twice a day, 21 days as a cycle.
  Interventions: Drug: TQB3006 tablets

INTERVENTIONS:
Drug: TQB3006 tablets — TQB3006 is an inhibitor protein.

SUMMARY:
This study includes two stage: dose escalation and dose extension, with a single dose and a multiple dose study. This is a single-center, open, non-randomized, single arm, study to evaluate the safety, tolerability and pharmacokinetics of TQB3006 tables in patients with advanced malignant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Age: 18 to 75 years old; an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Has at least one assessable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1;
* Female patient had no plans to become pregnant and voluntarily took effective contraceptive measures during the study period to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* There were other malignant tumors within 3 years;
* Has multiple factors affecting oral medication;
* Unalleviated toxicity ≥ grade 1 of CTCAE v5.0 due to any previous therapy , excluding hair loss;
* Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study，or have not fully recovered from previous surgery, or are expected to require major surgical surgery during the study period;
* Arteriovenous thrombotic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
* Have a history of psychotropic drug abuse and can not quit or have mental disorders;
* Subjects with any severe and / or uncontrolled disease including active hepatitis, a history of immunodeficiency, etc.;
* Tumor-related symptoms and treatment:

  1. Has known symptomatic central nervous system metastases and/or cancerous meningitis;
  2. Thoracic/abdominal/pericardial effusion with clinical symptoms or requiring repeated drainage, or drainage for the purpose of receiving treatment within 1 month after receiving the investigational drug for the first time;
  3. Has participated in other clinical trials within 4 weeks before first dose.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | At the end of Cycle 1 (21 Days).
  DLT will be defined as toxicities that meet pre-defined severity criteria (according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version5.0), and assessed as having a suspected relationship to study drug that occurred from first medication to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (21 Days).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended phase II dose (RP2D) | Baseline up to 24 months.
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3006 tablets in adult patients with Advanced Malignant Cancer

SECONDARY OUTCOMES:
Adverse events (AE) | 30 days after the last dose.
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | 30 days after the last dose.
  The occurrence of all serious adverse events (SAE).
Time to reach maximum plasma concentration (Tmax) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB3006 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Peak concentration (Cmax) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  The maximum observed plasma concentration of study drug. Each cycle is 21 days.
Half-life (t1/2) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Area under the concentration-time curve (AUC [0-infinity]) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  Area under the concentration-time curve from zero to infinity
Area under the concentration-time curve (AUC [0-t]) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  Area under the concentration-time curve from the first dose to a certain time point.
Apparent clearance (CL/F) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent volume of distribution (Vd/F) | Day 1: pre-dose, at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after-dose. Cycle 1 Day 1,Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day 21: pre-dose, Cycle 1 Day 21: at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after-dose. Each cycle is 21 days.
  Apparent volume of distribution of the TQB3006 in plasma.
Objective response rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  Defined as the percentage of patients with complete response (CR) or partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Chongqing university Cancer Hospital, Chongqing, Chongqing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan